CLINICAL TRIAL: NCT01491360
Title: Evaluation of the Safety & Efficacy of the LaserACE® Procedure to Restore Visual Function and Range of Accommodation
Brief Title: LaserACE® Procedure Restore Visual Function and Range of Accommodation LaserACE® Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ACE Vision Group, Inc. (Industry)
Collaborators: Vision Renu Taiwan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVG-2013-01
Record Dates: First submitted 2011-11-22; First posted 2011-12-14 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Presbyopia
Keywords: Presbyopia; sclera; LaserACE
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LaserACE(R) procedure performed (Experimental): The LaserACE(R) procedure (partial depth scleral micro-excisions with an Er:YAG laser in a specified pattern) will be performed.
  Interventions: Procedure: LaserACE(R)

INTERVENTIONS:
Procedure: LaserACE(R) — Partial depth scleral micro-excisions with an Er:YAG laser in a predetermined pattern.
  Other Names: LaserACE

SUMMARY:
A new minimally invasive procedure for treating presbyopia is being evaluated to determine if there is improvement in near and intermediate vision after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to understand and sign an informed consent;
2. Willing and able to attend postoperative examinations per protocol schedule;
3. 40 years of age or greater, of either gender or any race;
4. Less than (<) 1.00D of astigmatism in each eye, measured in their manifest refraction;
5. Mean refractive spherical equivalent refraction (MRSE) of +/- 0.50D for distance vision; Note: Subjects who meet this criterion as a result of prior laser refractive surgery (LASIK, LASEK or PRK) may qualify; however, the subject must have had the LVC procedure performed at least 12 months prior to the LaserACE® procedure and be stable.
6. Uncorrected distance visual acuity (UDVA) is better than or equal to 20/40 (logMAR 0.30) in each eye, and a Corrected Distance Visual Acuity (CDVA) is better than or equal to 20/32 (logMAR 0.20) in each eye;
7. Demonstrate Stereopsis of 200 seconds of arc or better using a Randot stereoscopic fly test and reading correction;
8. In good ocular health with the exception of presbyopia;
9. Presbyopia as demonstrated by:

   1. Currently wearing reading glasses and/or bifocals with an ADD of +1.50D or more; and
   2. Reduced near visual acuity when corrected for distance (DCNVA of 20/50 (logMAR 0.40) or worse; and
   3. Amplitude of accommodation (AA) of 1.50D or less as measured by the minus lens test; OR
   4. Amplitude of accommodation (AA) of 1.50D or less as measured by the iTrace aberrometer.
10. Intraocular pressure (IOP) >11mmHg and < 30 mmHg in each eye without IOP-lowering medication;
11. Less than or equal to (≤) 0.50D difference between the manifest refraction and the cycloplegic refraction;
12. Stable distance refraction is present, defined as ≤ 0.50D variation of refraction in the 12 months prior to the LaserACE® procedure. Manifest refraction cannot vary more than 0.50D from current spectacles that are at least 12 months of age, or from a documented refraction at least 12 months prior to the preoperative baseline exam;
13. Completed a washout period of two weeks (14 days) prior to LaserACE® procedure from prior treatment with:

    * NSAIDS, blood thinners, aspirin, and other substances which may increase bleeding;
    * Any anti-oxidant supplements (e.g., Vitamin B6, Vitamin B12, Vitamin E, Vitamin C, Acai, Ocuvite, etc);
    * Anti-oxidant food supplements, such as shitake mushroom, mushroom extract and oral anti-oxidants.

Exclusion Criteria

1. Self-reported current pregnancy or breast-feeding, or plans to become pregnant during the entire study period;
2. History of ocular trauma or prior ocular surgery, or expected to require retinal laser treatment or other ocular surgical intervention;
3. Presence of ocular pathology other than cataract such as:

   * Amblyopia or strabismus
   * Corneal abnormalities or disease
   * Dry Eye (International Task Force Level 3 or greater)
   * Pupil abnormalities (e.g., corectopia, Adie's)
   * Capsule or zonnular abnormalities
   * Intraocular inflammation
   * Retinal disease or pathology
   * Glaucoma (any type)
   * History of prior ocular surgery other than keratorefractive surgery;
4. Known pathology that may affect visual acuity and/or are predicted to cause future acuity losses to a level of 20/30 (logMAR 0.18) or worse (e.g., macular degeneration);
5. Previous radial keratotomy or other corneal surgery (e.g., corneal transplant, DSAEK/DSEK, lamellar keratoplasty), except for LASIK, EpiLASIK/LASEK, or PRK;
6. Previous anterior or posterior chamber surgery (e.g., vitrectomy, laser iridotomy);
7. Keratoconus or keratoconus suspect with CDVA of less than (<) 20/20 (< logMAR 0.00) at distance;
8. Near visual acuity at 40cm equivalent to their distance vision with distance correction (i.e., no evident effect of reduced accommodative range);
9. Use of systemic or ocular medications that may affect vision (the use of any miotic or cycloplegic agent is specifically contraindicated);
10. Acute or chronic disease or illness that could increase the operative risk or confound the study outcome(s) (e.g., diabetes mellitus, immunocompromised, connective tissue disease);
11. Uncontrolled systemic or ocular disease;
12. Any abnormality preventing reliable applanation tonometry in EITHER eye;
13. Undilatable pupil such that one cannot examine the periphery of the retina;
14. Functional eye preference, defined as phoria measuring over 15dp horizontally and/or over 2dp vertically, any strabismus, or suppression.
15. History of scleral ectasia, scleritis, or episcleritis; or thin sclera < 400 microns, as determined by taking the average of three measurements with ultrasound biomicroscopy (UBM) pachymetry;
16. History of nuclear sclerosis LOCS III grade 2 or worse and/or other cataracts reducing CDVA;
17. Known allergies to study medications including topical steroids, antibiotics and NSAIDS;
18. Per PI discretion

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with binocular near visual acuity of 20/32 (logMAR 0.20) or better at six months postoperatively with distance correction in place measured at 40cm and 60cm. | 6 months
  binocular near visual acuity of 20/32 (logMAR 0.20) or better at six months postoperatively with distance correction in place measured at 40cm and 60cm.

CONTACTS AND LOCATIONS:
Overall Officials: David Ma, MD, Principal Investigator — Chang Gung Memorial Hospital, Taipei, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hipsley A, Ma DH, Sun CC, Jackson MA, Goldberg D, Hall B. Visual outcomes 24 months after LaserACE. Eye Vis (Lond). 2017 Jun 16;4:15. doi: 10.1186/s40662-017-0081-y. eCollection 2017. PMID 28812042